CLINICAL TRIAL: NCT02533817
Title: Fructose and Ethnic Differences Study
Brief Title: Fructose and Ethnic Differences Study (FED Study)
Acronym: FED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BDM/12/13-7
Record Dates: First submitted 2015-07-30; First posted 2015-08-27 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: Fructose; Insulin; Postprandial lipemia; Ambulatory blood pressure; Ethnicity
MeSH Terms: conditions — Insulin Resistance | interventions — Dietary Sugars

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Sugar - Fructose (Experimental): Each participant consumed 20% daily caloric requirement as fructose.
  Interventions: Dietary Supplement: Dietary sugar
- Dietary Sugar - Glucose (Active Comparator): Each participant consumed 20% daily caloric requirement as glucose.
  Interventions: Dietary Supplement: Dietary sugar

INTERVENTIONS:
Dietary Supplement: Dietary sugar — This study examined the effect of high intakes of fructose compared to high intakes of glucose in a randomized crossover design. The treatment was in replacement of 20% of the daily caloric requirements for either fructose or glucose for each individual.

SUMMARY:
In the UK, people of black West African and Caribbean's tend to have healthier blood cholesterol and blood fat levels, as well as lower incidence of heart disease/heart attack. But rates of heart disease are now rising in young African-American populations with diabetes, for the first time exceeding the rate in their white European-American peers. One possible culprit is the increasing consumption of fructose which can lead to high blood fat levels. Fructose is a natural sugar found in fruits and table sugar but is also used the food industry as an ingredient and sweetener. Because fructose intakes are lower in the UK than in North America we are studying the effect of fructose intake in UK black West African and Caribbean people, to understand if fructose intake is indeed a reason for these ethnic differences.

DETAILED DESCRIPTION:
The overall nature of this study is to conduct an investigation into the metabolic effects of acute high fructose versus high glucose feeding in people of Black African (BA) compared to age and BMI-matched control subjects of White-European (WE) origin . The research question of our study is: do people of BA metabolise fructose differently than people of WE when challenged with a high sugar diet? Therefore, our specific aims are to determine the following in both people of BA and WE consuming both high fructose and high glucose meals: 1) the postprandial pattern of blood insulin, glucose, triglyceride and cholesterol concentrations; 2) ambulatory blood pressure measures during the postprandial period and 4) postprandial and 0-24-hour fasted serum and red blood cell membrane cholesterol and non-cholesterol sterol concentrations.

Potential participants will attend the scheduled screening session where the requirements of participation will be described and the participants will be given an opportunity to ask any questions they may have. Those still willing to participate will sign the informed consent form before the screening assessment is performed. Screening will require a fasted blood sample to be taken as well as a brief questionnaire to ascertain ethnicity (self-declared), medications and health status. An assessment of weight, height and waist circumference will also be taken to confirm they meet the inclusion criteria. It is expected that the results of the screening blood sample will be available within 1-2 weeks. Those participants meeting the inclusion criteria will be contacted and scheduled for the first study visit. Those not meeting the criteria will be notified by their preferred means of contact, a copy of their results will be provided.

Prior to attending participants treatment order will be randomized. Participants will report to the Metabolic Research Unit (MRU) at 08.00 following an overnight fast. A catheter will be inserted into an antecubital vein for collection of blood samples and a baseline blood sample collected at this time. Participant will be asked to undertake minimal physical activity during the remainder of the study period. A breakfast meal will be given at 0min, the lunch meal at 240min and meals will be consumed within 15 minutes. Participants will be fitted with a portable continuous blood pressure and heart rate monitor (arteriograph) and instructed on what to expect as it functions. Further blood samples will be taken at -30, -15, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 420min and at 24hrs (1440min, fasted). The energy content of the meals will be the estimated energy requirements of the participant (to the nearest 100kcals), with 20% of total daily energy coming from glucose or fructose. The glucose or fructose will be given dissolved water with added colour and orange/fruit flavours and provided at breakfast, lunch and supper. The remaining daily caloric requirement for each participant will be given a standardized evening meal to take away and consume at home.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported healthy, confirmed by blood tests (i.e. liver enzymes, full blood count, lipids, glucose); ethnicity White European participants had at least 3 grandparents originating from countries of Europe and Black African participants had at least 3 grandparents originating primarily from countries of West Africa (Economic Community of West African States (ECOWAS) and central African countries (e.g. Cameroon, Uganda, etc).

Exclusion Criteria:

* fasting glucose in the diabetic range (fasting glucose >7 mmol/l); hypertension (medically diagnosed or >140/90 mm Hg at screening); hyperlipidaemia deemed to require immediate medical intervention (defined as: total cholesterol >6.0 mmol/l; LDL-cholesterol >4.5 mmol/l; fasting TG >3 mmol/l).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Postprandial triglyceride concentrations | 0-420 minutes
  At time 0 minutes participants were provided with a study breakfast which they were required to consume within a 15 minute period and subsequent blood samples were drawn at 15, 30, 45, 60, 90, 120, 180, 240, 300, 360 and 420 minutes. The lunch meal was consumed immediately following the 240 minute blood sample and final fructose/glucose drink was consumed immediately following the 420 minute blood sample. A final blood sample was drawn at 24 hours under fasting conditions.

SECONDARY OUTCOMES:
Postprandial glucose concentrations. | 0-420 minutes
  At time 0 minutes participants were provided with a study breakfast which they were required to consume within a 15 minute period and subsequent blood samples were drawn at 15, 30, 45, 60, 90, 120, 180, 240, 300, 360 and 420 minutes. The lunch meal was consumed immediately following the 240 minute blood sample and final fructose/glucose drink was consumed immediately following the 420 minute blood sample. A final blood sample was drawn at 24 hours under fasting conditions.
Serum and red blood cell cholesterol and non-cholesterol sterol concentrations | 0 and 24-hour post treatment
  Blood samples collected at 0 and 24 hours post treatment consumption for serum and red blood cell membrane cholesterol and non-cholesterol sterol concentrations.
Postprandial insulin concentrations | 0-420 minutes
  At time 0 minutes participants were provided with a study breakfast which they were required to consume within a 15 minute period and subsequent blood samples were drawn at 15, 30, 45, 60, 90, 120, 180, 240, 300, 360 and 420 minutes. The lunch meal was consumed immediately following the 240 minute blood sample and final fructose/glucose drink was consumed immediately following the 420 minute blood sample.
Postprandial c-peptide concentrations | 0-420 minutes
  At time 0 minutes participants were provided with a study breakfast which they were required to consume within a 15 minute period and subsequent blood samples were drawn at 15, 30, 45, 60, 90, 120, 180, 240, 300, 360 and 420 minutes. The lunch meal was consumed immediately following the 240 minute blood sample and final fructose/glucose drink was consumed immediately following the 420 minute blood sample.
Postprandial non-esterified fatty acid concentrations | 0-420 minutes
  At time 0 minutes participants were provided with a study breakfast which they were required to consume within a 15 minute period and subsequent blood samples were drawn at 15, 30, 45, 60, 90, 120, 180, 240, 300, 360 and 420 minutes. The lunch meal was consumed immediately following the 240 minute blood sample and final fructose/glucose drink was consumed immediately following the 420 minute blood sample.

OTHER OUTCOMES:
Ambulatory blood pressure | Blood pressure was measured every 20 minutes during the postprandial period.
Serum uric acid concentrations | Serum uric acid concentrations measured at 0, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360 and 420 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Scott V Harding, PhD, Principal Investigator — King's College London

REFERENCES:
- [Derived] Goff LM, Whyte MB, Samuel M, Harding SV. Significantly greater triglyceridemia in Black African compared to White European men following high added fructose and glucose feeding: a randomized crossover trial. Lipids Health Dis. 2016 Sep 2;15(1):145. doi: 10.1186/s12944-016-0315-3. PMID 27590876